CLINICAL TRIAL: NCT03391674
Title: Fecal Microbiota Transplantation for Eradication of Carbapenem-resistant Enterobacteriaceae Colonization: A Randomized Control Trial
Brief Title: Fecal Microbiota Transplantation for Eradication of Carbapenem-resistant Enterobacteriaceae Colonization
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in protocol and delay in study initiation led to new study submission
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0338-19-RMB
Record Dates: First submitted 2017-12-04; First posted 2018-01-05 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Antibiotic Resistant Strain; Microbial Colonization
MeSH Terms: conditions — Communicable Diseases | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal Microbiota Transplantation (Experimental): Patients able to swallow will be given capsulized FMT using 15 capsules a day for two consecutive days. Patients will be treated concomitantly with omeprazole 20mg once in the evening before FMT and daily for the next 2 days.
  Interventions: Other: Fecal Microbiota Transplantation
- Observational (No Intervention): Observational

INTERVENTIONS:
Other: Fecal Microbiota Transplantation — Fecal Microbiota Transplantation through oral capsules after omeprazole pre-treatment
  Arms: Fecal Microbiota Transplantation

SUMMARY:
Antibiotic resistance has emerged world wide and is of major concern. Multidrug resistant (MDR) bacteria is widely spread and is now a major factor in morbidity and mortality in health-care settings. Among MDRs, carbapenem resistant Enterobacteriaceae (CRE) are of special concern, receiving the highest classification of "urgent threat level" in the US President Report. Consistent mortality rates of 40-50% are observed among inpatients with infections caused by CRE in hospitals worldwide, related mainly to unavailable, delayed or ineffective antibiotic treatment options. The extremely high mortality rates of patients with CRE infections have driven efforts to prevent the acquisition and spread of these bacteria in hospitals. These include screening for carriage, contact isolation of carriers, cohorting, dedicated healthcare staff and other infection control measures. These strategies have been proven as effective but are cumbersome and expensive. In most locations these strategies failed to completely eradicate CRE endemicity. CRE decolonization (eradication of colonization) might offer a double benefit - reducing the risk for the individual carrier to develop an infection due to the resistant strain (by that, potentially lowering the mortality risk) and preventing the bacteria from spreading to other patients, exposing them to the same hazard. Fecal microbiota transplantation (FMT), in which fecal material enriched with commensal microorganisms is transferred from a healthy donor, have proven efficacy in the treatment of recurrent Clostridium difficile infection (CDI) in multiple trails. Major adverse events that has been reported so far are mostly related to the route of administration (aspiration during nasogastric tube administration/colonoscopy). Other adverse events include mostly GI related symptoms (diarrhea, nausea, belching) and are self limited and resolve in few hours. FMT seems to be safe and effective both in immunocompetent and immunocompromised patients. The high efficacy of FMT in the treatment of a multi-drug resistant pathogen such as Clostridium difficile, suggest that it might be an efficient tool for other MDR pathogens (e.g. CRE). This study aim to assess the effects of FMT on colonization and clinical infections with CRE. The potential of FMT to restore the gut microbiome and compete with residual resistant strains offer a novel way to fight the current MDR epidemic. FMT will be applied in a randomized open label fashion to CRE carriers in a single center in Israel and will be given by capsules for 2 consecutive days followed by rectal sampling at predefined timepoint in the following 6 months.

DETAILED DESCRIPTION:
Antibiotic resistance has emerged world wide and is of major concern. Multidrug resistant (MDR) bacteria is widely spread and is now a major factor in morbidity and mortality in health-care settings. Among MDRs, carbapenem resistant Enterobacteriaceae (CRE) are of special concern, receiving the highest classification of "urgent threat level" in the US President Report. Consistent mortality rates of 40-50% are observed among inpatients with infections caused by CRE in hospitals worldwide, related mainly to unavailable, delayed or ineffective antibiotic treatment options. The extremely high mortality rates of patients with CRE infections have driven efforts to prevent the acquisition and spread of these bacteria in hospitals. These include screening for carriage, contact isolation of carriers, cohorting, dedicated healthcare staff and other infection control measures. These strategies have been proven as effective but are cumbersome and expensive. In most locations these strategies failed to completely eradicate CRE endemicity. CRE decolonization (eradication of colonization) might offer a double benefit - reducing the risk for the individual carrier to develop an infection due to the resistant strain (by that, potentially lowering the mortality risk) and preventing the bacteria from spreading to other patients, exposing them to the same hazard. Fecal microbiota transplantation (FMT), in which fecal material enriched with commensal microorganisms is transferred from a healthy donor, have proven efficacy in the treatment of recurrent Clostridium difficile infection (CDI) in multiple trails. Major adverse events that has been reported so far are mostly related to the route of administration (aspiration during nasogastric tube administration/colonoscopy). Other adverse events include mostly GI related symptoms (diarrhea, nausea, belching) and are self limited and resolve in few hours. FMT seems to be safe and effective both in immunocompetent and immunocompromised patients. The high efficacy of FMT in the treatment of a multi-drug resistant pathogen such as Clostridium difficile, suggest that it might be an efficient tool for other MDR pathogens (e.g. CRE). We aim to assess the effects of FMT on colonization and clinical infections with CRE. The potential of FMT to restore the gut microbiome and compete with residual resistant strains offer a novel way to fight the current MDR epidemic. FMT will be applied in a randomized open label fashion to CRE carriers in a single center in Israel and will be given by capsules for 2 consecutive days followed by rectal sampling at predefined timepoint in the following 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult inpatients ≥18 years positive for CRE of any strain and resistance mechanism in rectal surveillance stool samples, with or without CRE clinical samples. Positive rectal swab within one week before randomization will be mandatory.

Exclusion Criteria:

* Pregnant women
* Patients with severe neutropenia (<100/μl)
* Major abdominal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
CRE Decolonization defined as 3 consecutive negative rectal samples for CRE | 3 months after intervention
  3 consecutive negative rectal samples for CRE, last of which include a negative Polymerase chain reaction (PCR) test

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No